CLINICAL TRIAL: NCT05602545
Title: Comparison of Consumption of Some Fermented Foods and Nutrient Intakes in Individuals with Periodontal Disease and Periodontal Health
Brief Title: Periodontal Status in Fermented Food and Food Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuğba ŞAHİN (Other)
Responsible Party: Sponsor-Investigator, Tuğba ŞAHİN, Assistant professor, Abant Izzet Baysal University
Organization: Abant Izzet Baysal University (Other)
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: BAIBU-DH-TS-01
Record Dates: First submitted 2022-09-29; First posted 2022-11-02 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Periodontal Diseases
Keywords: fermented foods; periodontal health; periodontal disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Peri-implantitis (Experimental): patients with peri-implantitis
  Interventions: Other: food consumption in periodontal health and disease
- Peri-implant mucositis (Experimental): patients with peri-implant mucositis
  Interventions: Other: food consumption in periodontal health and disease
- Peri-implant health (Other): patients with peri-implant health
  Interventions: Other: food consumption in periodontal health and disease

INTERVENTIONS:
Other: food consumption in periodontal health and disease — To determine individuals' daily energy and nutrient intakes and the consumption amounts of food groups, food consumption records were kept by the nutritionist for three consecutive days, with one of them was weekend, using the 24-hour recall method. Data on individuals' frequency and amount of consumption of some fermented products were recorded, considering the foods available in our culture and the market.

SUMMARY:
Lack of certain nutrients and foods may negatively affect oral health. Therefore, nutrition plays an important role in maintaining oral health. This study aimed to evaluate and compare the nutrient intakes, consumption of food groups and some fermented foods of individuals with periodontal disease and health.

Ninety-three patients who applied to Periodontology Clinic were divided into three groups: periodontal health, gingivitis and periodontitis. In addition, plaque, gingival indices, bleeding on probing, periodontal pocket depth, and clinical attachment level were evaluated. To determine individuals' daily energy and nutrient intakes and the consumption amounts of food groups, food consumption records were kept by the nutritionist for three consecutive days, with one of them was weekend, using the 24-hour recall method. Data on individuals' frequency and amount of consumption of some fermented products were recorded, considering the foods available in our culture and the market.

ELIGIBILITY:
Inclusion Criteria:

* Patients with three teeth other than 20-year-old teeth in each jaw

Exclusion Criteria:

* Pregnancy and lactation,
* Patients with an acute oral lesion or necrotizing ulcerative periodontitis, -
* Patients with history of diabetes, rheumatic fever, lung and kidney disorders, and use of drugs that affect periodontal tissues (regular use of antibiotics, anti-inflammatory and mouthwashes),
* Patients who smoke, or patients who did not quit until last year were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
bleeding on probing | baseline
  To test for bleeding after probing, the probe is carefully introduced to the bottom of the pocket and gently moved laterally along the pocket wall. + is maximum and - is minimum.
periodontal pocket depth | baseline
  physical methods to measure the distance from the bottom of a pocket to a reference line, usually the gingival margin or the cemento-enamel junction.
Frequency of consumption of fermented foods | baseline
  the frequency of fermented foods is measured. The foods questioned were evaluated using a 7-point Likert-type frequency form (every day, 3-4 per week, 1-2 per week, 2 per month, 1 per month, never). In addition, the amounts of foods consumed each time were recorded, and the daily consumption amounts were obtained by dividing them by the frequency of consumption.
food consumption record | 1 or 3 days
  One or three days of consumption is recorded

SECONDARY OUTCOMES:
plaque index | baseline
  an index for estimating the status of oral hygiene by measuring dental plaque that occurs in the areas adjacent to the gingival margin. 0 is minimum and 3 is maximum. The situation worsens as the score increases.
gingival index | baseline
  The Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding. 0 is minimum and 3 is maximum. The situation worsens as the score increases.
clinical attachment level | baseline
  The clinical attachment level (CAL) and radiographically assessed bone levels are used to assess the loss of periodontal tissue support in periodontitis, a chronic, multifactorial inflammatory disease of the periodontium.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided